CLINICAL TRIAL: NCT00419198
Title: Postconditioning and Functional Recovery After Acute Myocardial Infarction
Brief Title: Clinical Outcomes of Angioplasty Postconditioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Michel Ovize, Pr., Hospices Civils de Lyon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2004.364
Record Dates: First submitted 2007-01-05; First posted 2007-01-08 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2010-03

CONDITIONS: Acute Myocardial Infarction
Keywords: Ischemia; Reperfusion; Myocardial infarction; Postconditioning
MeSH Terms: conditions — Ischemia; Myocardial Infarction | interventions — Ischemic Postconditioning

ARMS (2):
- 1 (Experimental): Post-conditioning during angioplasty
  Interventions: Procedure: Postconditioning
- 2 (Active Comparator): standard angioplasty
  Interventions: Procedure: standard angioplasty

INTERVENTIONS:
Procedure: Postconditioning — Postconditioning during angioplasty
  Arms: 1
Procedure: standard angioplasty — standard angioplasty without postconditioning
  Arms: 2

SUMMARY:
We previously demonstrated that postconditioning by coronary angioplasty can decrease infarct size (as measured by cardiac enzyme release) in patients with ongoing acute myocardial infarction. It is currently unknown whether postconditioning actually decreases or simply delays myocardial cell death during reperfusion. In addition, the long term effects of postconditioning on recovery of myocardial contraction remains elusive. The objective of the present study is to determine whether infarct size reduction by angioplasty postconditioning is maintained at 6 months and whether functional recovery is improved at one year post-infarction.

DETAILED DESCRIPTION:
Randomized, controlled, single-blinded trial comparing postconditioning to control (no intervention). Postconditioning consists of four episodes of one minute inflation followed by one minute deflation of the angioplasty balloon, starting within one minute of reflow after direct stenting of the occluded coronary artery.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, aged more than 18, with suspected first acute myocardial infarction, within 6 hours of the onset of chest pain, with a need for emergency revascularization by angioplasty. Patients must display a fully occluded (TIMI zero flow) culprit coronary artery, absence of visible collaterals and exhibit TIMI flow >2 after direct stenting by angioplasty.

Exclusion Criteria:

* Cardiac arrest or cardiogenic shock
* occlusion of the circumflex coronary artery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2005-09; Primary Completion 2008-03 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Infarct size as measured by cardiac enzymes and MRI at day 5 to 7 | during 72 hours after angioplasty, and at day 5 to 7

SECONDARY OUTCOMES:
Myocardial contraction (LV ejection fraction, wall motion score index, strain rate) measured by echocardiography at 6 month. | at 6 month

CONTACTS AND LOCATIONS:
Overall Officials: michel Ovize, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Michel Ovize, Lyon, France

REFERENCES:
- [Result] Thibault H, Piot C, Staat P, Bontemps L, Sportouch C, Rioufol G, Cung TT, Bonnefoy E, Angoulvant D, Aupetit JF, Finet G, Andre-Fouet X, Macia JC, Raczka F, Rossi R, Itti R, Kirkorian G, Derumeaux G, Ovize M. Long-term benefit of postconditioning. Circulation. 2008 Feb 26;117(8):1037-44. doi: 10.1161/CIRCULATIONAHA.107.729780. Epub 2008 Feb 11. PMID 18268150